CLINICAL TRIAL: NCT07301047
Title: App-Assisted Swallowing Program After Oral Cancer Surgery
Acronym: AASP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wenchuan Hsu, MS, nursing supervisor, Chang Gung Memorial Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202501330B0
Record Dates: First submitted 2025-12-09; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Oral Cancer; Reconstructive Surgery; Postoperative
Keywords: Oral Cancer; Postoperative; Reconstructive Surgery
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Intervention Model Description: This study adopts a quasi-experimental design using a non-randomized, two-group, pretest-posttest model. Participants are assigned sequentially to either the control or experimental group to avoid potential contamination between participants. The control group receives routine postoperative care, while the experimental group receives the same care plus an additional intervention using a swallowing exercise mobile application (App). Outcomes, including swallowing function, anxiety, and quality of life, are measured at baseline (pre-intervention), 4 weeks, and 12 weeks after surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swallowing Care + Exercise App Intervention (Experimental): Participants receive a swallowing care program combined with a mobile exercise App, starting on postoperative day 7. The App provides guided swallowing exercises, reminders, and progress tracking. Follow-up assessments at weeks 4 and 12.
  Interventions: Behavioral: Swallowing Care + Exercise App
- Routine Postoperative Care (Active Comparator): Participants receive standard postoperative care and routine ward education without the App-based swallowing intervention. Assessments at the same time points as the experimental group.
  Interventions: Behavioral: Routine Postoperative Care

INTERVENTIONS:
Behavioral: Swallowing Care + Exercise App — Participants receive a swallowing care program combined with a mobile exercise App, starting on postoperative day 7. The App provides guided swallowing exercises, reminders, and progress tracking. Follow-up assessments at weeks 4 and 12.
  Arms: Swallowing Care + Exercise App Intervention
Behavioral: Routine Postoperative Care — Participants receive standard postoperative care and routine ward education without the App-based swallowing intervention. Assessments at the same time points as the experimental group.
  Arms: Routine Postoperative Care

SUMMARY:
This study aims to examine the effects of a swallowing care program combined with an exercise mobile application (App) on swallowing function, anxiety, and quality of life in patients with oral cancer after flap reconstruction surgery. The goal is to determine whether integrating App-based swallowing exercises into postoperative care can improve rehabilitation outcomes compared with conventional care alone.

A purposive sampling method will be used to recruit 72 participants from the surgical wards of a medical center in northern Taiwan. Eligible patients scheduled for oral cancer tumor resection and flap reconstruction will be identified through consultation with plastic surgeons. After screening and informed consent, participants will be assigned to a control group or an experimental group, with approximately 36 patients in each group.

The control group will receive routine ward education and standard postoperative nursing care, while the experimental group will receive the same care plus an additional intervention using a swallowing exercise App. The intervention will begin on postoperative day 7, guided by the researcher. Follow-up assessments will be conducted during outpatient visits at postoperative week 4 and week 12. To minimize potential interference between participants, data collection will be performed sequentially-first for the control group, followed by the experimental group.

Data will be collected through self-administered questionnaires or researcher-assisted interviews, including a demographic survey, the Postoperative Oral Dysfunction-10 (POD-10), the Functional Oral Intake Scale (FOIS), a Visual Analog Scale for Anxiety, and the EORTC QLQ-H&N35 questionnaire for quality of life. Each assessment will take approximately 20-30 minutes. Participants may withdraw from the study at any time without penalty.

Descriptive statistics will be used to summarize participant characteristics. The chi-square test and independent t-test will be used to examine group homogeneity. Paired t-tests will be applied to evaluate within-group changes in swallowing function, anxiety, and quality of life before and after the intervention. The results of this study are expected to provide empirical evidence on the effectiveness of App-assisted swallowing rehabilitation for patients with oral cancer following reconstructive surgery, supporting the development of innovative, technology-based postoperative care models.

DETAILED DESCRIPTION:
This study adopts a purposive sampling method and will be conducted in surgical wards of a medical center in northern Taiwan. A total of 72 participants will be recruited, with approximately 36 patients in the experimental group and 36 in the control group, based on the sample size estimation.

Participants will be identified by the researcher through consultation with plastic surgeons regarding patients scheduled for oral cancer tumor resection and flap reconstruction surgery. Eligible patients will be screened according to inclusion and exclusion criteria. One day before surgery, the researcher will explain the study purpose and procedures to each patient. Those who agree to participate will sign an informed consent form and complete the baseline questionnaires either by self-administration or interview.

After surgery, when patients return to the ward, the intervention will begin on postoperative day 7. Participants will be divided into two groups:

Control group: receives routine ward education and standard postoperative care. Experimental group: receives the same routine care plus an additional intervention using a swallowing exercise mobile application (App). The researcher will assist participants in downloading and using the App.

Follow-up assessments will be conducted at 4 weeks and 12 weeks after surgery during outpatient clinic visits. To prevent contamination between participants, data will be collected sequentially-first from the control group and then from the experimental group.

Data collection instruments include a demographic questionnaire, the Postoperative Oral Dysfunction-10 (POD-10), Functional Oral Intake Scale (FOIS), Visual Analog Scale for Anxiety, and EORTC QLQ-H&N35 for quality of life. Each interview or questionnaire session will take approximately 20-30 minutes. Participants may withdraw at any time during the data collection process without penalty.

Data analysis will be performed using descriptive statistics to summarize participant characteristics. Homogeneity between groups will be tested using chi-square and independent t-tests. Paired t-tests will be used to compare pre- and post-intervention differences within groups. The study aims to evaluate the effects of an App-based swallowing exercise intervention on swallowing function, anxiety, and quality of life among patients with oral cancer after flap reconstruction surgery.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign a written informed consent form
* Diagnosed with oral cancer
* Hospitalized for first-time oral cancer tumor resection and flap reconstruction surgery
* Aged 18 years or older
* Conscious and mentally clear
* Able to communicate in Mandarin or Taiwanese

Exclusion Criteria:

* Diagnosed by a physician with poor postoperative wound healing that prevents participation in oral rehabilitation exercises
* Unable to perform oral rehabilitation exercises within one week after surgery, as determined by a physician

Withdrawal Criteria:

-Participants who withdraw consent at any time during the study will be excluded from further participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Oral Dysfunction-10 (POD-10) questionnaire | Beginning on postoperative day 7, and during outpatient visits at postoperative week 4 and week 12.
  Swallowing-related oral dysfunction was assessed using the Postoperative Oral Dysfunction-10 (POD-10) questionnaire. The POD-10 is a patient-reported outcome measure consisting of 10 items, with total scores ranging from 0 to 40, where higher scores indicate more severe oral dysfunction.
The Functional Oral Intake Scale (FOIS) | Beginning on postoperative day 7, and during outpatient visits at postoperative week 4 and week 12.
  Functional swallowing ability was evaluated using the Functional Oral Intake Scale (FOIS), a 7-point ordinal scale ranging from Level 1 (nothing by mouth) to Level 7 (total oral diet with no restrictions), where higher scores represent better oral intake function.

SECONDARY OUTCOMES:
anxiety | begin on postoperative day 7, during outpatient visits at postoperative week 4 and week 12.
  Anxiety levels were assessed using the Visual Analog Scale for Anxiety (VAS-A). The scale ranges from 0 to 10, where 0 indicates no anxiety and 10 indicates the highest level of anxiety, with higher scores reflecting greater anxiety severity.

OTHER OUTCOMES:
Change in Quality of Life Scores Measured by EORTC QLQ-H&N35 at 4 and 12 Weeks After Surgery | postoperative day 7, during outpatient visits at postoperative week 4 and week 12.
  Quality of life was assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Head and Neck 35 (EORTC QLQ-H&N35). The questionnaire comprises multiple head and neck cancer-specific symptom items, with scores linearly transformed to a 0-100 scale. Higher scores indicate greater symptom burden and poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Yean Hsiao Chiu, PHD, Study Director — Taipei Medical University
Locations (1):
- Chang Gung Memorial Hospital, Linkou Branch, Taoyuan District, Taoyuan City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Not applicable. Individual participant data will not be shared. Only aggregated study results may be published in scientific journals.

REFERENCES:
- See also: Chang Gung Memorial Hospital Official Website — https://www.cgmh.org.tw/
- Available data/document: No individual participant data (IPD) or supporting documents will be shared. Only aggregated study results may be published in journals or presented at conferences.: No individual participant data — https://www.cgmh.org.tw/ — No individual participant data (IPD) or supporting documents will be shared. Only aggregated study results may be published in journals or presented at conferences.